CLINICAL TRIAL: NCT01445756
Title: Topical Lidocaine for Pain Control With IUD Insertion: A Randomized Controlled Trial
Brief Title: Topical Lidocaine for Pain Control With Intrauterine Device (IUD) Insertion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-2010-0062
Record Dates: First submitted 2011-08-23; First posted 2011-10-04 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: Intrauterine Device
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Lidocaine (Active Comparator): Topical Lidocaine
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — During the procedure (placement of the IUD), 1ml of gel will be applied to the anterior lip of the cervix. After 1 minute of waiting, a tenaculum will be placed to steady the cervix. The catheter will be introduced into the cervical canal, past the external os and 1-1.5ml of gel will be placed into the canal. After another minute, the IUD will be placed in the standard fashion.
  Arms: Topical Lidocaine
Drug: Placebo — Placebo; no topical lidocaine administered
  Other Names: No intervention
  Arms: Placebo

SUMMARY:
Intrauterine contraception is a very effective, long term, reversible form of birth control, and is increasingly used in young, nulliparous patients. However, there is potential for pain with insertion of an Intrauterine Device (IUD) - particularly in patients without a previous history of vaginal delivery. The potential pain associated with insertion is often a significant barrier for patients when choosing and IUD for contraception. Several methods of pain control have been studied, but none have been shown to reduce pain at time of insertion. Our research question is to determine if 2% topical lidocaine gel, instilled into the cervical canal, will reduce maximum pain at time of insertion of a popular IUD (Mirena Intrauterine System) in young, nulliparous patients. This will be studied in a randomized, double-blind placebo-controlled trial.

DETAILED DESCRIPTION:
The investigators research question is to determine if 2% topical lidocaine gel, instilled into the cervical canal, will reduce maximum pain at time of insertion of a popular IUD (Mirena Intrauterine System) in young, nulliparous patients. This will be studied in a randomized, double-blind placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old

Exclusion Criteria:

* Age <18
* Non-English speaking
* Illiterate
* History of pregnancy with delivery >20 weeks
* History of prior IUD insertion or attempt

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in pain level from no Lidocaine administered to after Lidocaine is administered | Pain assessments prior to procedure, immediately after procedure, and 10 minutes after the procedure
  The investigators plan to engage 40 patients in this study, and will ask each to fill out a questionnaire that covers age, ethnicity, pregnancy history, reason for IUD insertion and recent medication use. Patients will be asked to assess their pain on 3 separate occasions during the visit, by marking an X on a Visual Analog Scale. Providers will also be asked to fill out a questionnaire covering their experience with the interventions as well as their assessment of the patients' pain during the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Landry, MD, Principal Investigator — University of Wisconsin Health Services
Locations (1):
- University Health Services Women's Care Clinic, Madison, Wisconsin, United States